CLINICAL TRIAL: NCT06174493
Title: Understanding Patient Engagement Trends in Atopic Dermatitis Clinical Research
Brief Title: Investigating Participation Patterns of Patients in Atopic Dermatitis Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 66783591
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials, specifically focused on atopic dermatitis, are crucial in assessing the safety and efficacy of new treatments. These trials serve as fundamental instruments in determining whether emerging medications outperform standard therapies, providing compelling evidence to support wider implementation.

The main goal is to thoroughly scrutinize trial completion rates and voluntary withdrawals among this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participant must be 18 years of age or older
* Confirmed diagnosis of atopic dermatitis

Exclusion Criteria:

* Enrolled in another research study
* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atopic dermatitis who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of atopic dermatitis patients who decide to enroll in a clinical research | 3 months
Rate of atopic dermatitis patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shalom G, Kridin K, Raviv KO, Freud T, Comaneshter D, Friedland R, Cohen AD, Ben-Amitai D. Atopic Dermatitis and Celiac Disease: A Cross-Sectional Study of 116,816 Patients. Am J Clin Dermatol. 2020 Feb;21(1):133-138. doi: 10.1007/s40257-019-00474-2. PMID 31679111
- [Background] Schut C, Dalgard FJ, Bewley A, Evers AWM, Gieler U, Lien L, Sampogna F, Stander S, Tomas-Aragones L, Vulink N, Finlay AY, Legat FJ, Titeca G, Jemec GB, Misery L, Szabo C, Grivcheva-Panovska V, Spillekom-van Koulil S, Balieva F, Szepietowski JC, Reich A, Roque Ferreira B, Lvov A, Romanov D, Marron SE, Gracia-Cazana T, Svensson A, Altunay IK, Thompson AR, Zeidler C, Kupfer J; ESDAP Study collaborators. Body dysmorphia in common skin diseases: results of an observational, cross-sectional multicentre study among dermatological outpatients in 17 European countries. Br J Dermatol. 2022 Jul;187(1):115-125. doi: 10.1111/bjd.21021. Epub 2022 May 22. PMID 35041211
- [Background] Patruno C, Fabbrocini G, Longo G, Argenziano G, Ferrucci SM, Stingeni L, Peris K, Ortoncelli M, Offidani A, Amoruso GF, Talamonti M, Girolomoni G, Grieco T, Iannone M, Nettis E, Foti C, Rongioletti F, Corazza M, Veneri MD, Napolitano M; Dupilumab for Atopic Dermatitis of the Elderly (DADE) Study Group. Effectiveness and Safety of Long-Term Dupilumab Treatment in Elderly Patients with Atopic Dermatitis: A Multicenter Real-Life Observational Study. Am J Clin Dermatol. 2021 Jul;22(4):581-586. doi: 10.1007/s40257-021-00597-5. PMID 33725337

DOCUMENTS (1):
  • Informed Consent Form (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06174493/ICF_000.pdf